CLINICAL TRIAL: NCT03356301
Title: Study of the Remodeling of the Ascending Aorta During the Sports Season in Long Distance Triathletes Versus Controls
Brief Title: Study of the Aorta Adaptations to Exercise in Triathletes During Sports Season (CoATri)
Acronym: CoATri
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-A01872-51
Record Dates: First submitted 2017-11-22; First posted 2017-11-29 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2019-01

CONDITIONS: Stiffness, Aortic; Cardiac Remodeling, Ventricular; Vascular Remodeling; Magnetic Resonance Imaging, Functional; Athletes
Keywords: Aortic compliance; Aortic distensibility; CMR; Triathletes; Ventriculo-atrial coupling
MeSH Terms: conditions — Ventricular Remodeling; Vascular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triathletes (Experimental): Every triathlete will realize three cardiac MRI exams.The second of those will be done at the fitness peak, 2-3 weeks before the main objective of the sports season. Training will be increased between the study beginning and the first MRI, and the second exam. After each cardiac MRI, an applanation tonometry examination will aslo be performed.
  Interventions: Device: Cardiac MRI; Device: Applanation tonometry
- Controls (Experimental): Every control subject will also realize three cardiac MRI exams if possible at the same time as the triathletes.They must be not engaged in physical activity more than 150 minutes a week on average. After each cardiac MRI, an applanation tonometry examination will aslo be performed.
  Interventions: Device: Cardiac MRI; Device: Applanation tonometry

INTERVENTIONS:
Device: Cardiac MRI — Non injected cardiac MRI exam
Device: Applanation tonometry — Applanation tonometry and ECG

SUMMARY:
Regular sustained physical activity creates a cardiac remodelling : it is athlete's heart. In our preliminary work published in 2016, the investigators demonstrated in a small population of triathletes that there is also a vascular remodelling named athlete's artery. Moreover, the investigators know that left ventricle and aorta behave together like a couple. So they want to study by Cardiovascular Magnetic Resonance Imaging the impact of triathlon on the cardiac AND aortic remodelling.

ELIGIBILITY:
Inclusion Criteria:

* to be enrolled in a social security plan.
* to have a BMI between 18,5 and 25 kg/m²
* to have received full information on the organization of the research and having signed its informed consent
* to have carried out a clinical screening adapted to the research

  *** Triathlete group:
* to have a minimum performance level: between 2h and 2h45 on an M triathlon during the past year (provide proof),
* to participate in 2018 in a long distance triathlon, i. e. at least distance L
* to have a defined training volume: less than 8 hours per week during the winter months and between 10 and 15 hours per week in preparation of the objective

  ***Control group:
* to have no more than 150 minutes of moderate physical activity per week (footing, brisk walking, cycling, etc.).

Exclusion Criteria:

* Persons referred to in Articles L. 1121-5 to L. 1121-8 and L1122-2 of the Public Health Code
* Cardiovascular history including Ii.e. known heart rhythm disorders
* Chronic disease: diabetes, high blood pressure...
* Long-term drug therapies that may modify cardiovascular remodeling such as Conversion Enzyme Inhibitor, Angiotensin II Receptor Antagonist,
* Active smoking, even if occasional
* Contraindication to MRI

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Aortic compliance in triathletes in mm2/mmHG | at baseline, at the fitness peak (6 to 10 months later) and at recovery (3 to 6 months after the fitness peak)
  aortic compliance = pulsed pressure-to-absolute variation of aortic surface ratio

CONTACTS AND LOCATIONS:
Overall Officials: Damien MANDRY, MD,PhD, Principal Investigator — CHRU de Nancy; Anne-Charlotte DUPONT, MD, Principal Investigator — CHRU de Nancy
Locations (1):
- Central Hospital, Nancy, France

REFERENCES:
- [Background] Dupont AC, Poussel M, Hossu G, Marie PY, Chenuel B, Felblinger J, Mandry D. Aortic compliance variation in long male distance triathletes: A new insight into the athlete's artery? J Sci Med Sport. 2017 Jun;20(6):539-542. doi: 10.1016/j.jsams.2016.10.009. Epub 2016 Oct 29. PMID 27838232